CLINICAL TRIAL: NCT01436630
Title: Comparação Entre o Teste de Caminhada de Seis Minutos e o Teste do Degrau de Seis Minutos em Pacientes Com Acidente Vascular Encefálico
Brief Title: Step Test and Six Minute Walk Test in Stroke
Status: Completed | Type: Observational
Sponsor: Faculdades Metropolitanas Unidas (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Comparação Entre o Teste de Caminhada de Seis Minutos e o Teste do Degrau de Seis Minutos em Pacientes Com Acidente Vascular Encefálico., Faculdades Metropolitanas Unidas
Other Study IDs: TDS-2809
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Stroke
Keywords: Exercise Tolerance; Step Test; Stroke; Walking
MeSH Terms: conditions — Stroke | interventions — Exercise Test; Walking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke: To accomplish the study it was assessed a group of 12 post-stroke patients who were admitted in the Rehabilitation Clinic inside the University. As inclusion criteria it was established to be able to walk alone without supervision and with no aids.
  All the patients signed an informed consent before performing the tests. To characterize the sample it were used the Fugl-Meyer scale, Orpington test, Mini Exam of the Mental State and some other data regarding the age, gender, type of the lesion and side of the lesion.
  Interventions: Other: Step Test and Six Minute Walk.

INTERVENTIONS:
Other: Step Test and Six Minute Walk. — The 6 Minute Walk Test (6MWT) was conducted in a level corridor 30 meters long and 5 meters wide. Before and after testing were measured O2 saturation (SatO2) and heart rate (HR), respiratory rate (RR), blood pressure (BP), the Double Product (DP), a measure of myocardial oxygen consumption, was calculated as the product of HR and systolic BP, and the sensation of dyspnea and fatigue of the lower limbs using the Borg scale, and performing the record turns traveled, each 30 meters is considered a covered back. To calculate the predicted distance, the investigators use the formula described by American Thoracic Society (ATS) knowing the weight, age and height of participants. The Step Test (ST) was conducted in six minutes for it to be compared to the 6MWT.
  Other Names: Step Test; Six Minute Walk Test

SUMMARY:
The purpose of this study is to investigate the viability of using the Step Test (ST) in stroke patients, and to compare the functional performance of the physiologic variables in stroke patients during ST and Six Minute Walk Test (6MWT).

DETAILED DESCRIPTION:
To accomplish the study it was assessed a group of 12 post-stroke patients who were admitted in the Rehabilitation Clinic inside the University. As inclusion criteria it was established to be able to walk alone without supervision and with no aids.

ELIGIBILITY:
Inclusion Criteria:

* To be able to walk alone without supervision and with no aids.

Exclusion Criteria:

* There were no.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-stroke patients
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Physiological Variables | 6 months
  Will be assessed Blood Pressure (BP), Heart Rate (HR), Breathing, Feeling of fatigue and dyspnea with the Borg scale, and the Double Product.

SECONDARY OUTCOMES:
Performance | 6 months
  Will be evaluated through the correlation between the number of ascents on the step and the distance covered in walking test.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Daminello Raimundo, Professor, Principal Investigator — Faculdades Metropolitanas Unidas; Camila Torriani-Pasin, Professor, Study Director — University of Sao Paulo; Carlos Bandeira de Mello Monteiro, Professor, Study Director — University of Sao Paulo; Osmar Aparecido Theodoro Junior, Professor, Study Director — Faculdades Metropolitanas Unidas; Talita Dias da Silva, Physiotherap, Study Chair — Faculdades Metropolitanas Unidas
Locations (1):
- Faculdades Metropolitanas Unidas, São Paulo, São Paulo, Brazil